CLINICAL TRIAL: NCT06942884
Title: Dexamethasone and Dexmedetomidine Versus Dexmedetomidine Alone With Bupivacaine in Ultrasound Guided Rectus Sheath Block in Midline Abdominal Surgeries
Brief Title: Dexamethasone and Dexmedetomidine Versus Dexmedetomidine Alone With Bupivacaine in Ultrasound Guided Rectus Sheath Block
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: sarah mohamed (Other)
Responsible Party: Sponsor-Investigator, sarah mohamed, lecturer, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 0108165
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Dexmedetomidine; Dexamethasone; Abdominal Surgeries
MeSH Terms: interventions — Dexmedetomidine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): Patients will receive bilateral RSB with 20 ml on each side containing 10 ml 0.5% bupivacaine, 20μg dexmedetomidine, 4mg dexamethasone and normal saline.
  Interventions: Drug: Dexmedetomidine and dexamethasone in addition to bupivacaine in rectus sheath block
- group 2 (Active Comparator): Patients will receive bilateral RSB with 20 ml on each side containing 10 ml 0.5 bupivacaine, with 4mg dexamethasone and normal saline
  Interventions: Drug: dexamethsone in addition to bupivacaine in rectus sheath block

INTERVENTIONS:
Drug: Dexmedetomidine and dexamethasone in addition to bupivacaine in rectus sheath block — addition of dexmedetomidine to dexamethasone in rectus sheath block
  Other Names: group 1
  Arms: group 1
Drug: dexamethsone in addition to bupivacaine in rectus sheath block — addition of dexamethasone in rectus sheath block
  Other Names: group 2
  Arms: group 2

SUMMARY:
Major abdominal surgery involves a variety of surgical procedures on a variety of patients, necessitating a broad spectrum of pain and analgesic needs.

A crucial element of multimodal analgesia that spares the use of opioids is regional anaesthesia.

Rectus sheath block (RSB) is a common regional block for post-operative analgesia after abdominal surgeries with midline incisions. A good analgesic effect has been reported for upper as well as lower abdominal midline incisions.(2) It was firstly described in 1899 with the aim of deposition of local anaesthetic (LA) in the virtual space between the posterior wall of the rectus abdominis muscle and its sheath. The anaesthetic injected into this space is proposed to spread freely up and down to block the anterior branches of the thoracoabdominal nerves before they emerge from the rectus sheath. The ventral branches of the lower thoracic nerves (T6-T12), which are located between the rectus abdominis muscle and its sheath, innervate the central region of the anterior abdominal wall.

In general, a single injection of local anesthetic can give analgesia for 4-12 hours following surgery, depending on the drug's chemical composition and degree of lipid solubility. Since postoperative pain might last for several days, prolonging the duration of action of local anaesthetics is important.(5) To prolong the postoperative analgesic period of local anaesthetics, many adjuncts have been used, including fentanyl, neostigmine, clonidine, and most recently dexamethasone and dexmedetomidine.(6) Dexamethasone is a highly potent, long-acting glucocorticoid. It reduces the activity of nociceptive C-fibres via binding to glucocorticoid receptors, which inhibits potassium conductance. It may also lengthen the duration of analgesia by systemic anti-inflammatory actions and local vasoconstrictive action.

Dexmedetomidine is one of the α -adrenoceptor agonists with α2 -adrenoceptor selectivity with both analgesic and sedative properties. it shortens the duration of the sensory and motor blockade while lengthening the initial blocking time when used as a perineural adjuvant

DETAILED DESCRIPTION:
AIM OF THE WORK The aim of the current study is to compare between adding dexamethasone with dexmedetomidine versus dexamethasone alone in ultrasound-guided RSB.

Primary aim:

The total amount of opioids used from completion of surgery till 48 hours.

Secondary aim:

The time to rescue analgesics need, duration of post operative analgesia, severity of postoperative pain at rest and with movement, the quality of recovery and any observed complications.

7. PATIENTS After approval of Local Ethics Committee and with written informed consent, this study will be conducted at Alexandria Main University Hospital and will be on 36 patients of both sexes, scheduled for major abdominal surgery.

Inclusion criteria

1. American Society of Anaesthesiologists (ASA) physical status I and II.
2. Patients aged 18-50 years.
3. Body mass index (BMI) less than 30 kg/m2.
4. Patients indicated for open abdominal surgeries with midline skin incision under general anaesthesia.
5. Elective and haemodynamically stable emergency cases. Exclusion criteria

1. Patients' refusal. 2. History of allergy to any of the study medications. 3. Diabetic patients. 4. Contraindications to regional anaesthesia, coagulopathy, anatomical abnormalities, haemodynamic instability, local infection, and suspected intra-abdominal sepsis.

8. METHODS

A- Preoperative assessment:

* Proper medical, surgical and drug history.
* General and airway examination.
* Laboratory investigations will be checked including:

Complete blood count (CBC), liver and kidney function tests and coagulation profile.

* Electrocardiography (ECG), and echocardiography (echo) for patients above 40 years.
* All patients will be informed about the study design, the analgesic regimen, and how to express pain intensity with the use of the VAS. The VAS is a 10-cm line corresponding to their pain level, with 0 at one end representing no pain at all and 10 at the other end representing the worst imaginable pain. Also the quality of recovery (QoR-15) (10) questionnaire will be illustrated.

B- Monitoring and patient preparation:

On arrival to the operating theater, an 18-G intravenous (IV) cannula will be inserted and IV Ringer's solution will be started according to the fluid chart of each patient.

Noninvasive blood pressure, pulse oximeter, and electrocardiography will be attached to the patients. Capnography will be attached with induction of general anesthesia.

C- Anaesthetic technique:

General anaesthesia with endotracheal intubation will be induced with 1 μg/kg fentanyl, 2 mg/kg propofol, and 0.5 mg/kg atracurium. Anaesthesia was 9. maintained with 1.2% isoflurane in 50% O2 in air mixture; additional boluses of 0.5-1 μg/kg fentanyl and 0.1 mg/kg atracurium will be given every 30 min until the end of the operation.

After completion of surgery, bilateral RSB will be performed under real-time ultrasound guidance (USG) using an in-plane approach. Under sterile precautions, the rectus sheath was identified at its lateral border, and a high-frequency linear probe is placed transversely across the linea semilunaris at or just above the level of the umbilicus. The lateral border of the rectus sheath is identified by the transition from the triple layer of muscle (external oblique, internal oblique, and transversus abdominis) on the lateral side to the single layer of muscle (rectus abdominis) medially. A 22-G needle will be inserted, the needle tip will be identified in-plane approach, and 20 ml of solution will be administered in the fascial plane between the rectus abdominis muscle and posterior wall of the rectus sheath, which is confirmed by hydrodissection under USG guidance.(11)

The 40 patients will be divided into two groups; each group includes 20 patients in double blinded study:

Group 1: Patients will receive bilateral RSB with 20 ml on each side containing 10 ml 0.5% bupivacaine, 20μg dexmedetomidine, 4mg dexamethasone and normal saline.

Group 2: Patients will receive bilateral RSB with 20 ml on each side containing 10 ml 0.5 bupivacaine, with 4mg dexamethasone and normal saline.

After completion of the analgesic intervention, a reversal agent was administered for neuromuscular recovery, and the patient will be extubated and shifted to the recovery room.

10. MEASUREMENTS

1. Demographic data (Age, Sex, BMI, Type of surgery). 2. The total amount of opioids used from completion of surgery till 48 hours. 3. The time to rescue analgesics need. 4. Duration of post-operative analgesia: Time from completion of the block to the first request of rescue analgesia.

5. The severity of post-operative pain at rest: Assessed using the VAS upon arrival to the PACU, after 30 and 60 min. The VAS was then recorded at 2, 4, 6, 8, 12, 24, 30, and 36 post-operative hours. Pain severity was categorized as mild (VAS≤3), moderate (3 ˂ VAS ˂ 7), and severe (VAS≥7).

6. The severity of post-operative pain with movement (bilateral knee flexion): Assessed using the VAS upon arrival to the PACU, after 30 and 60 min. The VAS was then recorded at 2, 4, 6, 8, 12, 24, 30, and 36 post-operative hours.

7. The quality of recovery by QoR-15 questionnaire: scores for excellent, good, moderate, and poor recovery were 136-150, 122-135, 90-121, and 0-89, respectively.(12) It is done before surgery as a baseline and after 24 hours.

8. Observed complications such as: bleeding, penetration of peritoneum or local anaesthetic toxicity.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists (ASA) physical status I and II.
* Patients aged 18-50 years.
* Body mass index (BMI) less than 30 kg/m2.
* Patients indicated for open abdominal surgeries with midline skin incision under general anaesthesia.
* Elective and haemodynamically stable emergency cases.

Exclusion Criteria:

* Patients' refusal.
* History of allergy to any of the study medications.
* Diabetic patients.
* Contraindications to regional anaesthesia, coagulopathy, anatomical abnormalities, haemodynamic instability, local infection, and suspected intra-abdominal sepsis.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
postoperative opioid consumption | postoperative day 2
  mg

SECONDARY OUTCOMES:
postoperative pain score | postoperative day 2
  0 no pain to 10 sever pain
quality of recovery 15 | postoperative day 2
  0-150
complications | postoperative day 2
  bleeding , local anesthetic toxicity

CONTACTS AND LOCATIONS:
Overall Officials: sarah m elgamal, MD, Principal Investigator — Alexandria University
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pirie K, Traer E, Finniss D, Myles PS, Riedel B. Current approaches to acute postoperative pain management after major abdominal surgery: a narrative review and future directions. Br J Anaesth. 2022 Sep;129(3):378-393. doi: 10.1016/j.bja.2022.05.029. Epub 2022 Jul 6. PMID 35803751